CLINICAL TRIAL: NCT02967666
Title: Evaluation of PET/MRI Using a Somatostatin Analog Tracer as a Novel Approach to Detecting Pathology in High Risk TB-exposed Contacts
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOTANOC_contacts
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — 68Ga-DOTANOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG PET/MRI, DOTANOC PET/MRI (Experimental): FDG PET/MRI and DOTANOC PET/MRI will be performed.
  Interventions: Radiation: FDG ligand; Radiation: DOTANOC ligand

INTERVENTIONS:
Radiation: FDG ligand
  Other Names: 18F-Fludeoxyglucose
Radiation: DOTANOC ligand
  Other Names: 68Ga-DOTANOC

SUMMARY:
PET/MRI (positron emission tomography/magnetic resonance imaging) with somatostatin analog tracers has the potential to provide an imaging technique targeting subclinical granulomatous disease in those with latent tuberculosis (TB), allowing identification of individuals who may be at risk of progression to active TB.

DETAILED DESCRIPTION:
Granulomas, the hallmark of TB infection, have an increased density of somatostatin receptors. Somatostatin analog PET tracers, such as 68Ga-DOTANOC, bind to somatostatin receptors and are able to detect pulmonary TB lesions using PET/MRI. This study aims to better understand the pathology of the spectrum of latent TB using 68Ga-DOTANOC PET/MRI imaging, identifying individuals with subclinical pulmonary TB who may be at risk of progressing to active TB.

Currently, biomarkers to identify those who are at risk of developing active TB are limited. Non-invasive biomarkers for pulmonary lesions are sorely needed and imaging with 68Ga-DOTANOC PET/MRI provides an opportunity to detect subclinical pulmonary disease in those who have been in close contact with smear-positive pulmonary TB.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or over
2. Close household contact of any patient with newly-diagnosed (within last 2 months) smear positive pulmonary TB (close contact defined as sleeping in the same house for at least one month with a TB patient prior to start of treatment).
3. Interferon Gamma Release Assay (IGRA) positive
4. Willing to comply with the study visits and procedures
5. Willing and able to provide written informed consent

Exclusion Criteria:

1. Previous treatment for TB disease
2. Diabetes that is, in the judgment of the investigator, so poorly controlled that it would prevent adequate PET scanning
3. Cardiac pacemaker, aneurysm clip or other metallic implant considered unsafe for MRI
4. Occupation involving substantial exposure to radiation
5. Malignancy requiring chemotherapy or radiation
6. Known lung disease which may affect interpretation of the scan
7. Known chronic kidney disease
8. Symptoms, signs and/or previous investigations suggestive of active TB in the opinion of the investigator (cough for >1 month, cough productive of sputum or blood, shortness of breath, weight loss, night sweats, fever, abnormal examination, chest X-ray findings)
9. Women who are currently pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) of 68Ga-DOTANOC in subclinical TB using PET/MRI | Within 2 months of exposure to smear-positive pulmonary TB

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore